CLINICAL TRIAL: NCT02619474
Title: The Effect of Whiteboards on Patient Satisfaction: A Prospective Controlled Study in BC's Children's Hospital
Brief Title: The Effect of Whiteboards on Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Seear, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H15-01896
Record Dates: First submitted 2015-10-19; First posted 2015-12-02 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Satisfaction; Physician-Patient Relations; Communication; Nurse-patient Relations
Keywords: Parent Satisfaction; Patient Satisfaction; Whiteboard; Communication
MeSH Terms: conditions — Personal Satisfaction; Communication; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Patients who have been admitted to the 3F or 3M wards under the care of the clinical teaching unit (CTU) after the introduction of the new, labelled whiteboard.
  Interventions: Other: Whiteboard
- Control (No Intervention): Patients who have been admitted to the 3R surgical ward under the care of any of the nursing groups without the introduction of the new labelled whiteboard.

INTERVENTIONS:
Other: Whiteboard — 1. On morning rounds, the child's management will be discussed with the family and the day's plan for treatment and investigations will be written on the whiteboard.
  2. The second step will be to review and update the whiteboard at the end of the day. Anything that has been left out or uncompleted will be highlighted and brought up on the following morning's rounds. Next, the nurse will ask the family to write down any questions.
  3. Lastly, on the afternoon before a child's discharge, the nurse will take particular care to make sure the parents write down all of their concerns prior to going home. These specific questions concerning discharge planning will be addressed in detail at rounds the following morning.
  Arms: Experimental

SUMMARY:
These days, particularly over the last decade, attention is being paid to the opinion of the patient and, in the case of pediatrics, the patient's family. Unfortunately, recent work has shown that this remains an imperfect process. Studies of inpatient families show that parents often leave hospital with only a minimal idea of side effects of drugs, who they can contact in the event that something goes wrong, and even something as simple as the date of the next medical visit. In fact, some studies have shown that adult patients don't even know the name of their doctor or nurse.

While there are several papers examining the degree of unhappiness of parents in hospitals, there is very little research looking at what can be done to improve a patient's sense of satisfaction with care (and communication) while in the hospital. One suggestion has been the provision of whiteboards in the room that can allow the family to have a better idea of what is going on during the child's day. These have been suggested but never exposed to prospective, quantitative study.

With the intention of improving the management of patients in the new Acute Care Centre, the department of strategic planning at Children's Hospital organized a three day IMPROVE session moderated by PHSA specialists in quality control. During this meeting, the clinical course of a child on the medical and surgical wards was mapped out. This allowed the group to examine various ideas aimed at improving the care of children passing through the hospital and the sense of parental satisfaction with the whole process.

The main conclusion from the meeting (based both on available literature and the clinical experience of the group), was that communication between the medical team and parents should be improved. It was also concluded that the best way to do this would be to have a regularly updated whiteboard in each room. Prior to starting this, it was generally felt that the introduction of whiteboards should be tested in a prospective controlled manner - starting with a baseline study of patient satisfaction.

DETAILED DESCRIPTION:
Initial quality control study.

Study design.

After discussion with senior nurses, residents, and physicians in the hospital, it was agreed that a baseline quality control study of patient satisfaction would be carried out on the medical and surgical wards. A UBC summer student was hired to administer the surveys. The initial stage of the study consisted of administering a previously validated questionnaire to families on the morning of their day of discharge. Families on the medical CTU and also surgical families were included. All information was obtained by face to face interview. No data was obtained from data bases or postal questionnaire.

Inpatient questionnaire. The questionnaire was developed by the health services research unit from the University of Oxford and has subsequently been used in Canadian hospitals. The questionnaire contains eight sub-headings that cover different aspects of the admission (courtesy, communication, comfort etc). Within each sub-heading there are five questions, each is scored from 1 (poor) to 4 (excellent). The result is eight separate sub-scores, each with a maximum of 20 points, plus a total score of 160 points.

Results.

Over 3 months, 150 families were enrolled from the medical and surgical wards. No parents refused to enter the study. The results are summarized in graph 1. The pattern of responses in the surgical and medical patients was surprisingly similar. In general, parents are satisfied with their care at Children's Hospital but, as graph 1 shows, there were two obvious areas for improvement. The first was simple communication between health care staff and the parents. The second, and more serious problem, was dissatisfaction with the discharge process (labelled as continuity on the graph).

Proposed prospective study of whiteboards.

The hospital's Inpatient Model of Care committee reviewed these findings and developed a protocol aimed at improving both communication and discharge planning. Fortunately, there has been considerable interest in the results of the first study. As a result, there is enthusiastic support for the second stage investigation of whiteboards. Nursing and medical staff have been very supportive and helpful. The introduction of this new protocol will be studied in a prospective controlled manner - this plan forms the basis of this ethics application. The details of the study are as follows:

Study Patients:

The patient groups will be the same ones used in the initial quality control study. The intervention group will be medical CTU patients. The control group will be surgical patients. There has been full support from medical and nursing staff in both areas. All rooms in the hospital already have whiteboards but they are rarely used except to collect fluid balance data. The study will examine the effects of a formalized use of whiteboards on rounds in the medical wards. In the surgical wards the whiteboards are used on an occasion basis. There will be no change to the usual surgical ward round routine.

Study protocol:

The first step has been to add standardized headings to the boards. This has already been completed. Apart from the patient's name and target date of discharge, the board includes details of the care team such as, doctor, nurse, and social worker. At the bottom of the board there is a space for family questions, and then next to that is a space for the day's plan.

The improved communication framework will consist of the following:

1. On morning rounds, the child's management will be discussed with the family and the day's plan for treatment and investigations will be written on the whiteboard.
2. The second step will be to update the whiteboard at the end of the day. The nursing team are fully engaged with this part of the study. The child's bed side nurse will sit with the family in the afternoon and review the day's plan. Anything that has been left out or uncompleted will be highlighted and brought up on the following morning's rounds. Next, the nurse will ask the family to write down any questions. These will be listed on the board and will be a priority to be discussed at rounds.
3. Lastly, on the afternoon before a child's discharge, the nurse will take particular care to make sure the parents write down all of their concerns prior to going home. These specific questions concerning discharge planning will be addressed in detail at rounds the following morning.

There will be no changes made to the usual ward routine for control patients on the surgical ward. There will be no other investigations associated with the study. In particular, there will be no laboratory or radiological investigations.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were admitted to the pediatric wards

Exclusion Criteria:

* Any patients/parents who do not wish to enroll in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Parent satisfaction as measured on questionnaire | 6 Months
  The questionnaire was developed by the health services research unit from the University of Oxford and has subsequently been used in Canadian hospitals. The questionnaire contains eight sub-headings that cover different aspects of the admission (courtesy, communication, comfort etc). Within each sub-heading there are five questions, each is scored from 1 (poor) to 4 (excellent). The result is eight separate sub-scores, each with a maximum of 20 points, plus a total score of 160 points.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Seear, MD, Principal Investigator — British Columbia's Children's Hospital
Locations (1):
- BC's Children's Hospital, Vancouver, British Columbia, Canada